CLINICAL TRIAL: NCT02051660
Title: German Randomized Controlled Trial of the Psychotherapeutic Intervention for Advanced Cancer Patients: Managing Cancer and Living Meaningfully (CALM)
Brief Title: German Evaluation of the Effectiveness of the Psychological Intervention Managing Cancer and Living Meaningfully (CALM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Collaborators: German Cancer Aid (Other); University of Hamburg-Eppendorf (Other); University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Anja Mehnert, Prof. Dr. Anja Mehnert, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DKH-110746; DKH-109967 (Other Grant/Funding Number: German Cancer Aid)
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Depression; Psychological Distress
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Manualized CALM Intervention (Experimental)
  Interventions: Behavioral: Manualized CALM intervention
- Non-manualized supportive intervention (Active Comparator)
  Interventions: Behavioral: Non-manualized supportive intervention.

INTERVENTIONS:
Behavioral: Manualized CALM intervention — Managing Cancer and Living Meaning Cancer (CALM) is a short-term individual psychotherapy for patients with advanced disease.
  Other Names: Managing Cancer and Living Meaning Cancer (CALM)
  Arms: Manualized CALM Intervention
Behavioral: Non-manualized supportive intervention. — Supportive psycho-oncological intervention.
  Arms: Non-manualized supportive intervention

SUMMARY:
Purpose of this randomized controlled trial is to test the efficacy of the individual psychotherapeutic intervention Managing Cancer and Living Meaningfully (CALM) in a German sample of patients with advanced cancer. The interventions aim is to reduce depression and distress and support psychological well-being.

DETAILED DESCRIPTION:
Principal hypothesis: The manualized psychotherapeutic intervention (CALM) will result in a significantly greater reduction in depression and psychological distress compared to a non-manualized supportive psycho-oncological intervention. Secondary hypothesis: The manualized psychotherapeutic intervention (CALM) will further result in a significantly improve psychological well-being, quality of life and sense of meaning compared to a non-manualized supportive psycho-oncological intervention.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Fluency in German
* No cognitive impairment indicated in the medical record or by the attending oncologist
* Confirmed diagnosis of solid tumors with UICC (Union Internationale Contre le Cancer) stages III/IV/ metastasized cancer (all with expected survival of 12-18 months)
* PHQ-9 depression score >=9 or Distress thermometer score >=5

Exclusion Criteria:

* Major communication difficulties (including language barriers)
* Inability to commit to the required 3-6 psychotherapy sessions
* A score <20 on the Short Orientation-Memory-Concentration (SOMC) test, indicating cognitive impairment unless deemed suitable at recruiter's discretion
* A score <70 on the Karnofsky-Performance Status Scale, indicating high physical symptom burden impeding study participation
* Being in psychotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Depression module of the Patient Health Questionnaire (PHQ-9) | 6-months
  A reliable and valid 9-item measure of depression.
Beck Depression-Inventory II (BDI-II) | 6-months
  A reliable and valid 21-item self-report instrument for evaluating the severity of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Anja Mehnert, Prof Dr, Principal Investigator — University Medical Center of Leipzig; Martin Härter, Prof Dr Dr, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (2):
- Germany (2):
  - Department of Medical Psychology and Medical Sociology, University Medical Center Leipzig, Leipzig, Saxony
  - Department of Medical Psychology, University Medical Center Hamburg-Eppendorf, Hamburg

REFERENCES:
- [Derived] Scheffold K, Philipp R, Vehling S, Koranyi S, Engelmann D, Schulz-Kindermann F, Harter M, Mehnert-Theuerkauf A. Spiritual well-being mediates the association between attachment insecurity and psychological distress in advanced cancer patients. Support Care Cancer. 2019 Nov;27(11):4317-4325. doi: 10.1007/s00520-019-04744-x. Epub 2019 Mar 18. PMID 30887126
- [Derived] Scheffold K, Philipp R, Engelmann D, Schulz-Kindermann F, Rosenberger C, Oechsle K, Harter M, Wegscheider K, Lordick F, Lo C, Hales S, Rodin G, Mehnert A. Efficacy of a brief manualized intervention Managing Cancer and Living Meaningfully (CALM) adapted to German cancer care settings: study protocol for a randomized controlled trial. BMC Cancer. 2015 Aug 19;15:592. doi: 10.1186/s12885-015-1589-y. PMID 26286128